CLINICAL TRIAL: NCT02527187
Title: Extract Allergen From Betula Verrucosa. Test Sensitivity and Specificity of Diagnostic in Prick Test Preparation.
Brief Title: Determination of the Sensitivity and Specificity of Prick Test Betula Verrucosa
Acronym: T502
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T502-SSP-007; 2013-005368-24 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Immune System Diseases
Keywords: Immune System Diseases; Prick Test; Betula verrucosa
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergic patients to birch pollen (Experimental): Allergic patients already diagnosed to be "true allergic" to birch pollen.
  A mean wheal diameter >3 mm obtained in a prick test with histamine dihydrochloride 10 mg/ml.Also presence of serum specific IgE and clinical history of symptomatology related to exposure to birch pollen.
  Patients of both gender aged from 5 up to 70 years.
  Interventions: Biological: 10 HEP/mL Betula verrucosa allergen extract; Biological: 25 HEP/mL Betula verrucosa allergen extract; Biological: 50 HEP/mL Betula verrucosa allergen extract; Biological: 100 HEP/mL Betula verrucosa allergen extract
- Non-allergic patients to birch pollen (Experimental): Patients already diagnosed to be "true non-allergic" to birch pollen.
  Non clinical history of symptomatology related to the exposure to birch pollen. Previous skin prick test negative and absence or undetectable serum specific IgE to Betula verrucosa
  Patients of both gender aged from 5 up to 70 years.
  Interventions: Biological: 10 HEP/mL Betula verrucosa allergen extract; Biological: 25 HEP/mL Betula verrucosa allergen extract; Biological: 50 HEP/mL Betula verrucosa allergen extract; Biological: 100 HEP/mL Betula verrucosa allergen extract

INTERVENTIONS:
Biological: 10 HEP/mL Betula verrucosa allergen extract — The investigational product contained 10 HEP/mL Betula verrucosa allergen extract and was tested by administration onto skin. The test was carried out on the forearm following prick test technique.
Biological: 25 HEP/mL Betula verrucosa allergen extract — The investigational product contained 25 HEP/mL Betula verrucosa allergen extract and was tested by administration onto skin. The test was carried out on the forearm following prick test technique.
Biological: 50 HEP/mL Betula verrucosa allergen extract — The investigational product contained 50 HEP/mL Betula verrucosa allergen extract and was tested by administration onto skin. The test was carried out on the forearm following prick test technique.
Biological: 100 HEP/mL Betula verrucosa allergen extract — The investigational product contained 100 HEP/mL Betula verrucosa allergen extract and was tested by administration onto skin. The test was carried out on the forearm following prick test technique.

SUMMARY:
The main objective is to evaluate the concentration of allergen extract of Betula verrucosa that elicit a papule equivalent to that produced by a solution of histamine dihydrochloride 10 mg / ml in size.

DETAILED DESCRIPTION:
Open, prospective, unblinded and non-randomized biological assay. Each patient was tested with four concentrations of allergen and with a histamine and saline solution as positive and negative controls, respectively.

ELIGIBILITY:
General inclusion criteria for both groups:

* Positive skin prick test with the positive control (Histamine HCl at 10 mg/mL). The length of the largest diameter of the wheal induced by this control should be ≥ 3 mm.
* Negative skin prick test with the negative control. The length of the largest diameter of the wheal induced by this control should be < 3 mm.
* All ages and both genders.

For the group of patients CH+ (true positive to Betula verrucosa): All these patients had a previous diagnosis of allergy to the birch pollen:

* A positive case history with inhalant allergy related to exposure to birch pollen.
* A positive skin prick test (mean wheal diameter ≥ 3 mm) when tested with a biologically standardized extract prepared from birch pollen. This preparation, from another manufacturer, was the one used in the routine in the Hospital.
* Positive test for specific IgE (CAP value > 0.35 IU/mL). For the group of patients CH- (true negative to Betula verrucosa): All these patients had a previous diagnosis of allergy to agents unrelated to birch pollen.
* A negative case history with inhalant allergy related to exposure to birch pollen or to pollen with known cross-reactivity with the birch pollen. These patients could be allergic to other pollen or other allergens, such mites.
* A negative prick test (largest diameter of the wheal ≥ 3 mm) when tested with a standardized extract prepared from the allergen source in question.
* A negative test for specific IgE (CAP value < 0.35 IU/mL) to birch pollen or to pollen with known cross-reactivity with birch pollen: Corylus avellana, Quercus verrucosa, Fagus sylvatica, Castanea satavia, Carpinus betelus and Alnus glutinosa.

Exclusion criteria for both groups:

* Patients that were using drugs that may interfere with the skin prick tests.
* Patients using the following drugs 24 hours before the test: theophylline, systemic corticosteroids.
* Patients in which the largest diameter of the wheal induced by the positive control was < 3 mm.
* Patients in which the largest diameter of the wheal induced by the negative control was ≥ 3 mm.
* Pregnancy, dermographism, atopic dermatitis (locally at the test site), urticaria.
* Patients who suffer disease in which the use of adrenaline is not allowed.
* Patients with any severe psychiatric disease.

For the patients CH+:

• Patients that received or are treated with immunotherapy with an allergenic extract of birch pollen and/or with allergen extracts with known cross-reactivity to birch pollen (Corylus avellana, Quercus verrucosa, Fagus sylvatica, Castanea satavia, Carpinus betelus and Alnus glutinosa).

For the patients CH-:

* Patients sensitized to pollen with demonstrated cross-reactivity with the pollen of Betula verrucosa. These pollen included Corylus avellana, Quercus verrucosa, Fagus sylvatica, Castanea satavia, Carpinus betelus and Alnus glutinosa.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Boquete, MD, Study Director
Locations (1):
- Hospital Lucus Augusti, Lugo, Galicia, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening based on subjects already diagnosed as allergic or not to birch pollen. (See Inclusion criteria section)
Period: Overall Study
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Started | 75 | 126
Completed | 75 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients were included for the analysis and tested with the 4 concentrations of the birch extract, negative and positive controls, and with the birch pollen extract used in normal clinical conditons Skin prick test was considered positive when wheal diameter was >3mm and negative when wheal diameter was < 3 mm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen | Total
Number analyzed (Participants) | 75 | 126 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 12 | 22
  Between 18 and 65 years | 60 | 104 | 164
  >=65 years | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (15.5) | 40.8 (14.3) | 39.8 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 80 | 122
  Male | 33 | 46 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 75 | 126 | 201
Region of Enrollment [Number; unit: participants]
  Spain | 75 | 126 | 201
positive skin prick test (diameter of the wheal > 3mm) [Count of Participants; unit: Participants] | 75 | 126 | 201

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity for 100 HEP/mL
Description: Sensitivity for 100 HEP/mL concentration of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of positives that are correctly identified by the test.
  Sensitivity: True positives/Total disease
Time Frame: 1 hour
Measure: Number; unit: positive reaction
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
positive reaction | 75 | 0

2. Primary Outcome: Sensitivity for 50 HEP/mL
Description: Sensitivity for 50 HEP/mL concentration of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of positives that are correctly identified by the test.
  Sensitivity: True positives/Total disease
Time Frame: 1 hour
Measure: Number; unit: positive reaction
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
positive reaction | 74 | 0

3. Primary Outcome: Sensitivity for 25 HEP/mL
Description: Sensitivity for 25 HEP/mL concentration of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of positives that are correctly identified by the test.
  Sensitivity: True positives/Total disease
Time Frame: 1 hour
Measure: Number; unit: positive reaction
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
positive reaction | 63 | 0

4. Primary Outcome: Sensitivity for 10 HEP/mL
Description: Sensitivity for 10 HEP/mL concentration of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of positives that are correctly identified by the test.
  Sensitivity: True positives/Total disease
Time Frame: 1 hour
Measure: Number; unit: positive reaction
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
positive reaction | 58 | 0

5. Primary Outcome: Specificity for 100 HEP/mL
Description: Specificity for 100 HEP/mL concentrations of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of negatives that are correctly identified by the test.
  Specificity: True negatives/Total no disease.
Time Frame: 1 hour
Measure: Number; unit: Negative response
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
Negative response | 0 | 126

6. Primary Outcome: Specificity for 50 HEP/mL
Description: Specificity for 50 HEP/mL concentrations of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of negatives that are correctly identified by the test.
  Specificity: True negatives/Total no disease.
Time Frame: 1 hour
Measure: Number; unit: Negative response
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
Negative response | 0 | 126

7. Primary Outcome: Specificity for 25 HEP/mL
Description: Specificity for 25 HEP/mL concentrations of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of negatives that are correctly identified by the test.
  Specificity: True negatives/Total no disease.
Time Frame: 1 hour
Measure: Number; unit: Negative response
Groups:
- Allergic Patients to Birch Pollen: Allergic patients already diagnosed to be "true allergic" to birch pollen.
  A mean wheal diameter >3 mm obtained in a prick test with histamine dihydrochloride 10 mg/ml.Also presence of serum specific IgE and clinical history of symptomatology related to exposure to birch pollen.
  Patients of both gender aged from 5 up to 70 years.
  The investigational product contained the allergen extract of the pollen of Betula verrucosa and will be tested by administration onto skin. The test will be carried out on the forearm following prick test technique.
- Non-allergic Patients to Birch Pollen: Patients already diagnosed to be "true non-allergic" to birch pollen.
  Non clinical history of symptomatology related to the exposure to birch pollen. Previous skin prick test negative and absence or undetectable serum specific IgE to Betula verrucosa
  Patients of both gender aged from 5 up to 70 years.
  The investigational product contained the allergen extract of the pollen of Betula verrucosa and will be tested by administration onto skin. The test will be carried out on the forearm following prick test technique.
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
Negative response | 12 | 126

8. Primary Outcome: Specificity for 10 HEP/mL
Description: Specificity for 10 HEP/mL concentrations of the pollen of Betula verrucosa allergen extract used in skin prick test.
  It is the proportion of negatives that are correctly identified by the test.
  Specificity: True negatives/Total no disease.
Time Frame: 1 hour
Measure: Number; unit: Negative response
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
Number analyzed (Participants) | 75 | 126
Negative response | 16 | 126

ADVERSE EVENTS:
Time Frame: Up to 1 hour after performing test and up to 5 days after release from the hospital.
Description: In terms of safety, although skin prick tests are safe and patients were already tested previously in the hospital, the investigator took special care in order to check for the presence of any unwanted reaction. Patients remained in the hospital facilities (around 30 min-1 hour after test) and were instructed to report, to the investigator, any adverse event occurring after leaving the hospital.
Arm/Group | Allergic Patients to Birch Pollen | Non-allergic Patients to Birch Pollen
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/126
Other Adverse Events (participants affected / at risk) | 0/75 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No